CLINICAL TRIAL: NCT02396758
Title: Study of the OPTtimum Duration of Acoustic Pulse ThromboLYSis ProcEdure in the Treatment of Acute Submassive Pulmonary Embolism
Brief Title: Optimum Duration of Acoustic Pulse Thrombolysis Procedure in Acute Pulmonary Embolism
Acronym: OPTALYSE PE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: EKOS Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EKOS-12; 2016-000502-11 (EudraCT Number)
Record Dates: First submitted 2015-03-10; First posted 2015-03-24 (Estimated); Results first posted 2021-03-02 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Embolism and Thrombosis
MeSH Terms: conditions — Pulmonary Embolism; Thrombosis | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- APT/2 Hours-r-tPA/2 mg/hr/Catheter (Experimental): A total of 4 or 8 mg r-tPA (as 2 mg/hour [hr]/catheter) will be delivered through Ekosonic® Endovascular Device (EKOS) ultrasonic infusion catheter for 2 hrs.
  Interventions: Device: Ekosonic® Endovascular Device ultrasonic infusion catheter; Biological: Recombinant tissue plasminogen activator
- APT/4 Hours-r-tPA/1 mg/hr/Catheter (Experimental): A total of 4 or 8 mg r-tPA (as 1 mg/hr/catheter) will be delivered through EKOS ultrasonic infusion catheter for 4 hrs.
  Interventions: Device: Ekosonic® Endovascular Device ultrasonic infusion catheter; Biological: Recombinant tissue plasminogen activator
- APT/6 Hours-r-tPA/1 mg/hr/Catheter (Experimental): A total of 6 or 12 mg r-tPA (as 1 mg/hr/catheter) will be delivered through EKOS ultrasonic infusion catheter for 6 hrs.
  Interventions: Device: Ekosonic® Endovascular Device ultrasonic infusion catheter; Biological: Recombinant tissue plasminogen activator
- APT/6 Hours-r-tPA/2 mg/hr/Catheter (Experimental): A total of 12 or 24 mg r-tPA (as 2 mg/hr/catheter) will be delivered through EKOS ultrasonic infusion catheter for 6 hrs.
  Interventions: Device: Ekosonic® Endovascular Device ultrasonic infusion catheter; Biological: Recombinant tissue plasminogen activator

INTERVENTIONS:
Device: Ekosonic® Endovascular Device ultrasonic infusion catheter — r-tPA will be administered via EKOS.
  Other Names: Acoustic Pulse Thrombolysis Procedure (APT Procedure); EKOS
Biological: Recombinant tissue plasminogen activator — Recombinant tissue plasminogen activator will be administered as per the dose and schedule specified in the arm.
  Other Names: r-tPA

SUMMARY:
The objective is to determine the optimum dose of thrombolytic and duration of the ultrasound procedure (together defined as the APT Procedure) as a treatment for acute submassive pulmonary embolism (PE). Symptomatic submassive PE are participants with acute (less than or equal to [≤]14 days) PE with normal systemic arterial blood pressure (greater than [>] 90 mmHg) and evidence of RV dysfunction (right ventricular to left ventricular diameter ratio, that is; RV/LV ratio greater than or equal to [≥] 0.9). Participants with submassive PE will be randomized to one of four APT treatment groups: ultrasound of 2 and 6 hours (hrs) with r-tPA 2 milligrams (mg)/hr/catheter and ultrasound 4 and 6 hours with r-tPA, 1 mg/hr/catheter. On 08 June 2016, randomization into treatment group 4 (APT/6 hours-r-tPA/2 mg/hr/catheter) was closed following a reported intracranial hemorrhage (ICH) and death in a study participant in this arm.

DETAILED DESCRIPTION:
This study is designed to investigate the lowest recombinant tissue plasminogen activator (r-tPA) dose-ultrasound treatment time required to achieve the same reductions in thrombus burden and associated improvement in physiologic parameters demonstrated in ULTIMA (EKOS 08 [NCT01166997]) and SEATTLE II (EKOS 09 [NCT01513759]). Results of this study are intended to inform the study design for further studies of the Acoustic Pulse Thrombolysis (APT) Procedure. Analysis of the first 100 evaluable participants in the United States study suggested a degree of equipoise between treatment groups 1, 2 and 3 of the protocol and therefore the sample size has been extended and additional sites in the United Kingdom (UK) National Health Service included, with a view to adding to the findings of the OPTALYSE study from sites in the UK and increasing the number of participants treated by treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female greater than or equal to (≥) 18 years of age and less than or equal to (≤) 75 years of age.
2. CTA evidence of proximal PE (filling defect in at least one main or lobar pulmonary artery).
3. PE symptom duration ≤14 days.
4. Submassive PE: RV/LV diameter ≥ 0.9 from CTA and hemodynamically stable. For Participants in UK Sites: Submassive PE: RV/LV diameter ≥ 0.9 from CTA, hemodynamically stable and an elevated biomarker.
5. Must be treated within 48 hours of diagnosis of PE by CTA.
6. Signed Informed consent obtained from subject or Legally Authorized Representative.

Exclusion Criteria:

1. Stroke or transient ischemic attack (TIA), head trauma, or other active intracranial or intraspinal disease within one year.
2. Recent (within one month) or active bleeding from a major organ.
3. Major surgery within seven days of screening for study enrollment.
4. Clinician deems the subject high-risk for catastrophic bleeding.
5. History of heparin-induced thrombocytopenia (HIT).
6. Catheter-based pharmacomechanical treatment for PE within 3 days of study enrollment.
7. Systolic blood pressure (SBP) less than 90 mm Hg and/or use of vasopressors.
8. Cardiac arrest (including pulseless electrical activity and asystole) requiring active cardiopulmonary resuscitation (CPR).
9. Evidence of irreversible neurological compromise.
10. Life expectancy < one year. For Participants in UK Sites: Life expectancy < one year or enrollment in hospice care.
11. Use of thrombolytics or glycoprotein IIb/IIIa antagonists within 3 days prior to inclusion in the study.
12. Out-of-Range Laboratory Values: Hematocrit < 30%, Platelets < 100 thousand/microliter (μL), International normalized ratio (INR) > 3.
13. Creatinine outside the normal range for the treating institution.
14. Participant is pregnant (positive pregnancy test; women of childbearing capacity must be tested) or breast feeding.
15. Active cancer (metastatic, progressive, or treated within the last 6 months). Exception: participants with non-melanoma primary skin cancers are eligible to participate in the study.
16. Known allergy, hypersensitivity, or thrombocytopenia from heparin, r-tPA, or iodinated contrast except for mild-moderate contrast allergies for which steroid pre-medication can be used.
17. History of any hematologic disease potentially involving abnormal platelet number or function.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2015-06-12 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Tapson, MD, Principal Investigator — Cedar Sinai, Los Angeles
Locations (21):
- United States (16):
  - Cedars Sinai, Beverly Hills, California
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Florida Hospital Tampa, Tampa, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - University Hospital, Augusta, Georgia
  - St. Vincent Medical Group, Indianapolis, Indiana
  - Jewish Hospital, Louisville, Kentucky
  - East Jefferson General Hospital, Metairie, Louisiana
  - Detroit Medical Center, Detroit, Michigan
  - Mount Carmel Health System, Columbus, Ohio
  - UPMC Hamot, Erie, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Methodist Sugarland Hospital, Richmond, Texas
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Providence Sacred Heart Medical Center, Spokane, Washington
- United Kingdom (5):
  - Royal Devon & Exeter Hospital, Exeter, England
  - Medway Maritime Hospital, Gillingham, England
  - Royal Free Hospital, London, England
  - St. Thomas Hospital, London, England
  - Ninewells Hospital, Dundee, Scotland

REFERENCES:
- [Background] Piazza G, Sterling KM, Tapson VF, Ouriel K, Sharp ASP, Liu PY, Goldhaber SZ. One-Year Echocardiographic, Functional, and Quality of Life Outcomes After Ultrasound-Facilitated Catheter-Based Fibrinolysis for Pulmonary Embolism. Circ Cardiovasc Interv. 2020 Aug;13(8):e009012. doi: 10.1161/CIRCINTERVENTIONS.120.009012. Epub 2020 Aug 6. PMID 32757658
- [Result] Tapson VF, Sterling K, Jones N, Elder M, Tripathy U, Brower J, Maholic RL, Ross CB, Natarajan K, Fong P, Greenspon L, Tamaddon H, Piracha AR, Engelhardt T, Katopodis J, Marques V, Sharp ASP, Piazza G, Goldhaber SZ. A Randomized Trial of the Optimum Duration of Acoustic Pulse Thrombolysis Procedure in Acute Intermediate-Risk Pulmonary Embolism: The OPTALYSE PE Trial. JACC Cardiovasc Interv. 2018 Jul 23;11(14):1401-1410. doi: 10.1016/j.jcin.2018.04.008. PMID 30025734

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 131 subjects were randomized (ITT population) and 129 were treated (safety population). Two subjects were randomized into the trial but were not treated. One subject was randomized but prior to initiation of therapy, it was discovered the subject had chronic PE and was ineligible. One subject was randomized but decompensated prior to the initiation of therapy and expired. Due to changes in the protocol, there were no subjects enrolled in the UK in Treatment Arm 4.
Period: Overall Study
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Started | 38 | 37 | 38 | 18
Completed | 26 | 31 | 34 | 13
Not Completed | 12 | 6 | 4 | 5
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1
Not completed — Lost to Follow-up | 8 | 5 | 3 | 3
Not completed — Death | 1 | 1 | 0 | 1
Not completed — Randomized but not treated | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Overall number of participants
Groups:
- Total: Total of all reporting groups
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter | Total
Number analyzed (Participants) | 38 | 37 | 38 | 18 | 131
Age, Continuous [Median (Standard Deviation); unit: years] | 56.0 (13.05) | 57.9 (13.03) | 57.9 (12.3) | 58.2 (14.0) | 57.4 (12.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 21 | 7 | 62
  Male | 22 | 19 | 17 | 11 | 69
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian, not of Hispanic origin | 24 | 24 | 27 | 11 | 86
  African American, not of Hispanic origin | 12 | 10 | 9 | 6 | 37
  Hispanic or Latino | 0 | 2 | 0 | 0 | 2
  Asian or Pacific Islander | 0 | 1 | 1 | 0 | 2
  Other | 2 | 0 | 1 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 28 | 18 | 101
  United Kingdom | 10 | 10 | 10 | 0 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Right Ventricle (RV) Diameter-to-Left Ventricle (LV) Diameter Ratio to 48 ± 6 Hours After the Start of the APT Procedure
Description: Change from baseline in RV/LV will be determined by computed tomographic angiography (CTA).
Time Frame: Change from Baseline to 48 hrs ± 6 hours
Population: ITT population included all randomized participants. Here, 'Number analyzed' signifies participants evaluable for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 38 | 37 | 38 | 18
ratio
  Baseline: number analyzed (Participants) | 36 | 37 | 36 | 18
  Baseline | 1.53 (0.38) | 1.47 (0.35) | 1.52 (0.39) | 1.51 (0.58)
  Change at 48 ± 6 hours: number analyzed (Participants) | 35 | 35 | 35 | 18
  Change at 48 ± 6 hours | -0.43 (0.35) | -0.37 (0.26) | -0.41 (0.31) | -0.48 (0.51)

2. Primary Outcome: Number of Participants With Major Bleeding Within 72 Hours After Initiating the APT Procedure
Description: Criteria for major bleeding events, as defined by the International Society on Thrombosis and Haemostasis (ISTH): 1. Fatal bleeding and/or; 2. Symptomatic bleeding in a critical area or organ (intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome) and/or; 3. Bleeding causing a fall in hemoglobin level of 20 grams/liter (g/L) or more, or leading to transfusion of two or more units of whole blood or red blood cells.
Time Frame: Day 3 (within 72 hours after initiating the APT procedure)
Population: Safety population included all enrolled participants for whom the APT procedure was initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 37 | 37 | 37 | 18
Participants | 0 | 2 | 1 | 2

3. Secondary Outcome: Percentage of Participants With Treatment Success of an APT Procedure
Description: Treatment success of an APT procedure will be assessed by an Adjudication Committee that is blinded to the participant's treatment. The criteria for treatment success are defined as follows: A decrease in RV/LV from baseline to 48 hours after the start of the procedure of at least 0.2; and no life-threatening adverse events related to PE or its treatment through 30 days after the start of the APT procedure.
Time Frame: From Baseline up to Day 30
Population: ITT population included all randomized participants. Here, 'Overall number of participants analyzed' signifies evaluable participants per clinical judgement of Adjudication Committee.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 23 | 25 | 26 | 18
Percentage of participants | 73.9 [53.5 to 87.5] | 68.0 [48.4 to 82.8] | 69.2 [50.0 to 83.5] | 61.6 [38.6 to 79.7]

4. Secondary Outcome: Change From Baseline in RV/LV at Days 0, 2, 30, 90, and 365, as Assessed by Echocardiograph.
Description: An echocardiogram was obtained at specified timepoints to evaluate RV/LV.
Time Frame: Baseline (Day -2 [within -48 hrs of APT start]), Day 0 (within 4 hours after APT end), Day 2 (48 [± 6] hrs of APT start), Day 30 (± 5 days), Day 90 (± 10 days) and Day 365 (± 14 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 38 | 37 | 38 | 18
Ratio
  Baseline: number analyzed (Participants) | 34 | 35 | 31 | 18
  Baseline | 1.19 (0.25) | 1.20 (0.23) | 1.13 (0.17) | 1.20 (0.35)
  Change at 48 hrs post-APT: number analyzed (Participants) | 31 | 32 | 29 | 18
  Change at 48 hrs post-APT | -0.23 (0.22) | -0.29 (0.25) | -0.17 (0.20) | -0.29 (0.32)
  Change at Day 30 post-APT: number analyzed (Participants) | 33 | 29 | 31 | 14
  Change at Day 30 post-APT | -0.38 (0.27) | -0.37 (0.23) | -0.30 (0.20) | -0.37 (0.39)
  Change at Day 90 follow-up: number analyzed (Participants) | 28 | 29 | 30 | 12
  Change at Day 90 follow-up | -0.41 (0.29) | -0.39 (0.23) | -0.31 (0.22) | -0.43 (0.41)
  Change at Day 365 follow-up: number analyzed (Participants) | 22 | 27 | 26 | 12
  Change at Day 365 follow-up | -0.44 (0.30) | -0.46 (0.24) | -0.35 (0.15) | -0.32 (0.13)

5. Secondary Outcome: Change From Baseline in Tricuspid Annular Plane Systolic Excursion (TAPSE) at Days 0, 2, 30, 90, and 365, as Assessed by Echocardiograph
Description: The extent of displacement of the tricuspid valves, termed as TAPSE was measured at specified timepoints using echocardiogram.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 38 | 37 | 38 | 18
Millimeters
  Baseline: number analyzed (Participants) | 33 | 33 | 28 | 18
  Baseline | 16.32 (5.06) | 17.20 (5.14) | 16.39 (5.36) | 18.02 (5.54)
  Change at 4 hrs post-APT: number analyzed (Participants) | 29 | 28 | 26 | 17
  Change at 4 hrs post-APT | 0.27 (6.09) | 0.79 (4.86) | 0.51 (4.68) | 2.17 (4.15)
  Change at 48 hrs post-APT: number analyzed (Participants) | 28 | 31 | 26 | 18
  Change at 48 hrs post-APT | 2.86 (4.56) | 1.75 (4.65) | 2.61 (4.82) | 3.34 (6.14)
  Change at Day 30 post-APT: number analyzed (Participants) | 29 | 28 | 27 | 12
  Change at Day 30 post-APT | 5.42 (5.59) | 5.39 (4.64) | 2.36 (4.75) | 2.26 (5.55)
  Change at Day 90 follow-up: number analyzed (Participants) | 27 | 28 | 26 | 11
  Change at Day 90 follow-up | 6.32 (5.64) | 3.69 (5.44) | 3.97 (6.29) | 2.07 (5.86)
  Change at Day 365 follow-up: number analyzed (Participants) | 21 | 25 | 23 | 11
  Change at Day 365 follow-up | 6.83 (5.88) | 5.22 (4.72) | 4.79 (5.97) | 3.50 (5.98)

6. Secondary Outcome: Change From Baseline in Estimated Right Ventricular Systolic Pressure (RVSP) at Days 0, 2, 30, 90, and 365, as Assessed by Echocardiograph
Description: RVSP was measured at specified timepoints using echocardiogram.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 38 | 37 | 38 | 18
Millimeters
  Baseline: number analyzed (Participants) | 27 | 29 | 22 | 16
  Baseline | 31.59 (14.89) | 36.64 (19.02) | 35.57 (16.32) | 25.75 (11.09)
  Change at 4 hrs post-APT: number analyzed (Participants) | 23 | 23 | 18 | 14
  Change at 4 hrs post-APT | -2.18 (13.04) | -10.87 (15.32) | -3.54 (14.23) | 2.13 (13.74)
  Change at 48 hrs post-APT: number analyzed (Participants) | 21 | 26 | 21 | 15
  Change at 48 hrs post-APT | 0.98 (9.36) | -5.35 (18.45) | -9.31 (10.53) | -7.80 (11.69)
  Change at Day 30 post-APT: number analyzed (Participants) | 24 | 22 | 21 | 12
  Change at Day 30 post-APT | -7.92 (11.69) | -13.84 (15.47) | -14.06 (15.41) | -4.86 (18.07)
  Change at Day 90 follow-up: number analyzed (Participants) | 21 | 19 | 18 | 11
  Change at Day 90 follow-up | -8.30 (15.38) | -15.60 (16.90) | -16.39 (24.18) | -7.08 (15.30)
  Change at Day 365 follow-up: number analyzed (Participants) | 15 | 16 | 17 | 10
  Change at Day 365 follow-up | -9.78 (12.79) | -12.87 (13.17) | -18.96 (12.23) | -7.16 (16.57)

7. Secondary Outcome: Percentage of Participants With Collapse of the Inferior Vena Cava (IVC) With Respiration at Days 0, 2, 30, 90, and 365, as Assessed by Echocardiograph
Description: The collapse of IVC was measured at specified timepoints using echocardiogram.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 38 | 37 | 38 | 18
percentage of participants
  Baseline: number analyzed (Participants) | 29 | 29 | 25 | 16
  Baseline | 96.55 [82.82 to 99.39] | 100.00 [88.30 to 100.00] | 96.00 [80.46 to 99.29] | 81.25 [56.99 to 93.41]
  4 hrs post-APT: number analyzed (Participants) | 29 | 25 | 28 | 16
  4 hrs post-APT | 89.66 [73.61 to 96.42] | 96.00 [80.46 to 99.29] | 89.29 [72.80 to 96.29] | 87.50 [63.98 to 96.50]
  48 hrs post-APT: number analyzed (Participants) | 24 | 31 | 28 | 17
  48 hrs post-APT | 100.00 [86.20 to 100.00] | 100.00 [88.97 to 100.00] | 92.86 [77.35 to 98.02] | 82.35 [58.97 to 93.81]
  Day 30 post-APT: number analyzed (Participants) | 29 | 27 | 30 | 13
  Day 30 post-APT | 96.55 [82.82 to 99.39] | 96.30 [81.72 to 99.34] | 96.67 [83.33 to 99.41] | 92.31 [66.69 to 98.63]
  Day 90 post-APT: number analyzed (Participants) | 25 | 25 | 28 | 12
  Day 90 post-APT | 100.00 [86.68 to 100.00] | 92.00 [75.03 to 97.78] | 96.43 [82.29 to 99.37] | 100.00 [75.75 to 100.00]
  Day 365 post-APT: number analyzed (Participants) | 18 | 23 | 23 | 12
  Day 365 post-APT | 94.44 [74.24 to 99.01] | 100.00 [85.69 to 100.00] | 86.96 [67.87 to 95.46] | 83.33 [55.20 to 95.30]

8. Secondary Outcome: Change From Baseline in Thrombus Burden by Miller Score as Assessed by Pulmonary Arteriogram (PAgram) at Day 0
Description: Miller score is composed of a score for arterial obstruction (objective score) and a score for reduction of peripheral perfusion of lungs (subjective evaluation). Right pulmonary artery (PA) is assigned 9 segmental arteries (3 to the upper, 2 to the middle, and 4 to the lower lobe), and left PA is assigned only 7 segmental arteries (2 to the upper, 2 to the lingula, and 3 to the lower lobe). Presence of segmental emboli, regardless of the degree of obstruction, is scored 1 point. Proximal emboli to the segmental level are scored a value equal to the number of segmental arteries arising distally. Maximal score of obstruction=16. Reduction of peripheral perfusion is scored by dividing each lung into upper, middle, and lower zones and by using a 4-point scale: 0=normal perfusion; 1=moderately reduced perfusion; 2=severely reduced perfusion; 3=no perfusion. Maximal score of reduced perfusion=18. Thus, the maximal Miller score =34. Higher Miller score=more thrombus burden.
Time Frame: Baseline, Day 0 (within 4 hours after APT end)
Population: ITT population included all randomized participants. Here, 'Overall number of participants analyzed' signifies participants with available pre and post PAgrams. 'Number analyzed' = participants evaluable for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 21 | 24 | 24 | 15
units on a scale
  Baseline | 23.71 (3.21) | 23.29 (6.00) | 24.21 (3.01) | 22.93 (2.99)
  Change at 4 hrs post-APT: number analyzed (Participants) | 4 | 7 | 9 | 5
  Change at 4 hrs post-APT | -1.00 (3.46) | -2.29 (5.62) | -3.11 (3.89) | -9.20 (3.11)

9. Secondary Outcome: Change From Baseline in Thrombus Burden by Modified Miller Score as Assessed by CTA Scan at 48 ± 6 Hours After the Start of the APT Procedure
Description: Modified miller score quantifies thrombus burden on CTA scans. Each segmental pulmonary artery (9 on the right, 7 on the left) that is fully or partly occluded by thrombus is given a score of 1. Any further proximal involves vessels score the number of segmental branches distal to that vessel, thereby giving a modified miller score of 0 (no thrombus) to 16 (thrombus in all segmental arteries or saddle embolism).
Time Frame: From Baseline to 48 hrs ± 6 hours
Population: ITT population included all randomized participants. Here, 'Number analyzed' signifies participants evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 38 | 37 | 38 | 18
units on a scale
  Baseline: number analyzed (Participants) | 36 | 37 | 36 | 18
  Baseline | 20.72 (2.76) | 20.00 (4.14) | 20.92 (2.31) | 20.44 (4.12)
  Change at 48 hrs post-APT: number analyzed (Participants) | 33 | 35 | 34 | 18
  Change at 48 hrs post-APT | -1.24 (1.71) | -2.20 (2.29) | -2.62 (2.47) | -5.22 (5.83)

10. Secondary Outcome: Change in 6 Minute Walk (6MW) Distance From Day 30 to Day 90 and 365
Description: The 6 minute Walk Test is a measure of functional exercise capacity. Participants will be asked to walk as far as possible within a 6-minute period, and the distance covered at the end will be noted and recorded.
Time Frame: Days 30, 90, 365
Population: ITT population included all randomized participants. Here, 'Number analyzed' signifies participants with evaluable data at specified timepoint.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 38 | 37 | 38 | 18
meters
  Day 30: number analyzed (Participants) | 28 | 30 | 35 | 9
  Day 30 | 355.4 (78.62) | 366.90 (157.76) | 362.3 (103.81) | 327.3 (99.70)
  Change at Day 90: number analyzed (Participants) | 24 | 28 | 34 | 8
  Change at Day 90 | 23.8 (133.98) | 70.6 (59.62) | 33.8 (65.85) | -6.3 (62.98)
  Change at Day 365: number analyzed (Participants) | 21 | 27 | 28 | 7
  Change at Day 365 | 21.6 (67.33) | 2.0 (175.11) | 57.9 (217.99) | -1.9 (155.78)

11. Secondary Outcome: Change in Borg Scale Score Before and After 6MW Distance Test at Days 30, 90, and 365
Description: Borg is a 10-point scale rating the maximum level of dyspnea (difficulty in breathing) and fatigue experienced before and after the 6MW distance test. Scores ranges from 0 (for no shortness of breath, or no fatigue) to 10 (for the greatest shortness of breath ever experienced, or maximum amount of fatigue felt). Higher scores indicates worse outcome.
Time Frame: Days 30, 90, and 365
Population: ITT population included all randomized participants. Here, 'Number analyzed' signifies participants evaluable for this outcome measure for specified categories
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 38 | 37 | 38 | 18
units on a scale
  Day 30: Dyspnea: number analyzed (Participants) | 28 | 30 | 35 | 10
  Day 30: Dyspnea | 0.75 [0 to 2] | 0 [0 to 2] | 0.5 [0 to 2] | 0 [0 to 2]
  Day 30: Fatigue: number analyzed (Participants) | 28 | 30 | 35 | 10
  Day 30: Fatigue | 0.25 [0 to 1.3] | 0 [0 to 0.5] | 0 [0 to 1] | 0 [0 to 0]
  Day 90: Dyspnea: number analyzed (Participants) | 26 | 30 | 36 | 10
  Day 90: Dyspnea | 1 [0 to 2] | 0.5 [0 to 1] | 0.5 [0 to 2] | 0 [0 to 3]
  Day 90: Fatigue: number analyzed (Participants) | 26 | 30 | 36 | 10
  Day 90: Fatigue | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 0.5] | 0 [0 to 0.5]
  Day 365: Dyspnea: number analyzed (Participants) | 22 | 27 | 30 | 10
  Day 365: Dyspnea | 0.25 [0 to 2] | 0.5 [0 to 1] | 0 [0 to 1] | 0 [0 to 3]
  Day 365: Fatigue: number analyzed (Participants) | 21 | 27 | 30 | 10
  Day 365: Fatigue | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 0]

12. Secondary Outcome: Number of Participants Who Received Oxygen Therapy
Description: Oxygen source is categorized as room air, nasal prongs, mask, and intubated.
Time Frame: Days 30, 90, and 365
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 38 | 37 | 38 | 18
Participants
  Day 30: Before 6MW test - Room air: number analyzed (Participants) | 29 | 30 | 34 | 10
  Day 30: Before 6MW test - Room air | 29 | 30 | 34 | 10
  Day 30: After 6MW test - Room air: number analyzed (Participants) | 28 | 30 | 33 | 10
  Day 30: After 6MW test - Room air | 28 | 30 | 33 | 10
  Day 90: Before 6MW test - Room air: number analyzed (Participants) | 26 | 30 | 36 | 10
  Day 90: Before 6MW test - Room air | 26 | 30 | 36 | 10
  Day 90: After 6MW test - Room air: number analyzed (Participants) | 26 | 30 | 36 | 10
  Day 90: After 6MW test - Room air | 26 | 30 | 36 | 10
  Day 365: Before 6MW test - Room air: number analyzed (Participants) | 21 | 27 | 30 | 10
  Day 365: Before 6MW test - Room air | 21 | 27 | 30 | 10
  Day 365: After 6MW test - Room air: number analyzed (Participants) | 21 | 28 | 30 | 10
  Day 365: After 6MW test - Room air | 21 | 28 | 30 | 10

13. Secondary Outcome: Change in Participant Reported Outcomes Measurement Information System Physical Function (PROMIS-PF) 6b Score From Day 30 to Day 365
Description: PROMIS-PF 6b questionnaire is developed by including 2-items from item-improved Health Assessment Questionnaire (HAQ) and 4-items from item-improved Physical Function-10 (PF-10) instruments. Both of these instruments assess participant's present abilities. Both "Item-Improved instruments" have 5-response options: HAQ - 1="without any difficulty," 2="with a little difficulty," 3="with some difficulty," 4="with much difficulty," 5="unable to do"; PF-10 - 1="not at all," 2="very little," 3="somewhat," 4="quite a lot," 5="cannot do." Total score is the average of all scores of component items, which ranges from 0 (no disability) to 100 (worst disability).
Time Frame: Day 30, Day 365
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 28 | 27 | 28 | 18
units on a scale
  Day 30: number analyzed (Participants) | 26 | 23 | 28 | 14
  Day 30 | 42.00 (10.905) | 43.86 (7.980) | 44.53 (6.695) | 41.40 (13.238)
  Change at Day 365: number analyzed (Participants) | 19 | 21 | 25 | 11
  Change at Day 365 | 3.61 (7.140) | 4.91 (8.909) | 2.14 (8.184) | 4.39 (8.699)

14. Secondary Outcome: Change in Pulmonary Embolism Quality of Life (PEmb-QOL) Score From Day 30 to Day 365
Description: The PEmb-QoL questionnaire contains 6 dimensions that has been created based on the contents of the items, frequency of complaints (Question [Q]1; score range: 1 [every day] to 5 [never]), activities of daily living (ADL) limitations (Q4; score range: 1 [limited a lot] to 3 [not at all]), work-related problems (Q5; response: yes/no), social limitations (Q6; score range: 1 [not at all] to 5 [extremely]), intensity of complaints (Q7 [pain in chest/shoulders]/8 [breathlessness]; score range: 1 [none] to 6 [very serious]) and emotional complaints (Q9; score range: 1 [at all times] to 6 [none of the times]). Total Score for all dimensions are calculated by the sum of the scores for each item of the dimension divided by the number of items. Total score ranges from 1 (better quality of life) to 100 (worst quality of life). Higher scores indicate poorer outcome (decreased quality of life). Questions 1, 4, 5, and 9 are reverse scored. Questions 2 and 3 provide descriptive information.
Time Frame: Day 30, Day 365
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 38 | 37 | 38 | 18
units on a scale
  Day 30: number analyzed (Participants) | 35 | 32 | 38 | 14
  Day 30 | 38.30 (25.723) | 27.85 (20.715) | 24.25 (18.109) | 25.63 (26.923)
  Change at Day 365: number analyzed (Participants) | 26 | 30 | 34 | 11
  Change at Day 365 | -16.79 (16.500) | -8.86 (26.576) | -8.75 (15.549) | -12.01 (14.832)

15. Secondary Outcome: Number of Participants Who Encountered Technical Procedural Complications
Description: Technical complications associated with the use of the EKOS device will be recorded during catheter placement in the pulmonary artery and during the infusion procedure.
Time Frame: From device placement through Day 2
Population: Safety population included all enrolled participants for whom the APT procedure was initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 37 | 37 | 37 | 18
Participants | 0 | 0 | 1 | 0

16. Secondary Outcome: Number of Participants With Symptomatic Recurrent Pulmonary Embolism (Per Adjudication)
Description: Number of participants with symptomatic recurrent pulmonary embolism up to 365 days following the APT procedure, were reported. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: From Baseline up to Day 365
Population: Safety population included all enrolled participants for whom the APT procedure was initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 37 | 37 | 37 | 18
Participants | 0 | 1 | 1 | 0

17. Secondary Outcome: Number of Participants Who Die Due to Any Cause
Description: Number of participants who died due to any cause for up to 365 days following the APT procedure, were reported.
Time Frame: From Baseline up to Day 365
Population: Safety population included all enrolled participants for whom the APT procedure was initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 37 | 37 | 37 | 18
Participants | 1 | 1 | 0 | 1

18. Secondary Outcome: For Participants of UK Sites: Freedom From Major Harm Occurring Between Enrolment and 30 Days
Description: Number of UK participants with freedom from major harms assessed by Safety Monitor using the following criteria: 1) Mortality - all cause and PE related; 2) Cardiovascular (CV) collapse defined as one or more of the following: a) Greater than (>) 40 millimeters of mercury (mmHg) drop in systolic blood pressure (SBP) (for >15 minutes from documented blood pressure as an in-patient) despite intravenous (IV) fluid challenge and absence of new atrial arrhythmia; b) Requirement for emergency systemic thrombolysis; c) Requirement for emergency surgical embolectomy ; d) Requirement for vasopressors; e)and/or Intubation/Ventilation; 3) Major bleeding per ISTH; 4) Recurrent PE (confirmed by imaging); and/or 5) Surgical correction of device related complication. Due to changes in the protocol, there were no subjects enrolled in the UK in Treatment Arm 4.
Time Frame: From Baseline up to Day 30
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 10 | 10 | 10 | 0
Participants | 10 | 9 | 9 | 0

19. Secondary Outcome: For Participants of UK Sites:Change in EuroQual - 5 Dimensions - 5 Levels (EQ-5D-5L) Score From Day 30 to Day 365
Description: The EQ-5D-5L consists of 2 parts - the descriptive system (Index Score) and the EQ Visual Analogue scale (VAS Score). The EQ-5D-5L descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression) and each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4), and extreme problems (5). Each one digit number expressing the level selected for each dimension is combined into a 5-digit number describing the respondent's heath state. These 5-digit numbers are converted into an index value, where 1 represents full health and 0 is equivalent to death. The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale with 100 being the best health imaginable and 0 being the worst health imaginable. Due to changes in the protocol, there were no subjects enrolled in the UK in Treatment Arm 4.
Time Frame: Day 30, Day 365
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 10 | 10 | 10 | 0
units on a scale
  Day 30 - EQ-5D-5L Index Score: number analyzed (Participants) | 8 | 9 | 10 | 0
  Day 30 - EQ-5D-5L Index Score | 0.732 (0.2624) | 0.819 (0.195) | 0.934 (0.134) |
  Day 30- EQ-5D-5L VAS Score: number analyzed (Participants) | 9 | 9 | 10 | 0
  Day 30- EQ-5D-5L VAS Score | 66.7 (19.04) | 77.8 (12.02) | 82.5 (7.91) |
  Change at Day 365 - EQ-5D-5L Index Score: number analyzed (Participants) | 6 | 9 | 9 | 0
  Change at Day 365 - EQ-5D-5L Index Score | 0.039 (0.0418) | -0.107 (0.252) | -0.042 (0.149) |
  Change at Day 365 - EQ-5D-5L VAS Score: number analyzed (Participants) | 7 | 9 | 9 | 0
  Change at Day 365 - EQ-5D-5L VAS Score | -1.6 (35.97) | -0.4 (22.01) | 7.1 (9.12) |

20. Secondary Outcome: For Participants of UK Sites: Time From Hospital Admission to Diagnosis of PE
Description: Duration of time between hospital admission and the diagnosis of pulmonary embolism (PE) measured in hours for UK participants.Due to changes in the protocol, there were no subjects enrolled in the UK in Treatment Arm 4.
Time Frame: From Baseline through Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 10 | 10 | 10 | 0
hour | 10.77 (10.78) | 9.30 (19.08) | 7.29 (9.64) |

21. Secondary Outcome: For Participants of UK Sites: Time From Diagnostic Computed Tomography (CT) Scan to Initiation of Treatment for PE
Description: Duration of time between Diagnostic Computed Tomography (CT) Scan to Initiation of Treatment for pulmonary embolism (PE) measured in hours for UK Participants. Due to changes in the protocol, there were no subjects enrolled in the UK in Treatment Arm 4.
Time Frame: From Baseline through Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 10 | 10 | 9 | 0
hour | 25.33 (12.58) | 24.53 (13.93) | 30.08 (18.42) |

22. Secondary Outcome: For Participants of UK Sites: Time in Each Level of Care (Level 0 and 1; Level 2; and/or Level 3) Through Discharge
Description: Levels are defined according to National Framework Document: Level 0 - normal acute ward care (patients whose needs can be met through normal ward care in an acute hospital), Level 1 - acute ward care, with additional advice and support from the critical care team (Patients at risk of their condition deteriorating, or those recently relocated from higher levels of care, whose needs can be met on an acute ward with additional advice from a critical care team), Level 2 - more detailed observation or intervention (requiring more detailed observation or intervention including support for a single failing organ system or post-operative care and those 'stepping down' from higher levels of care) and Level 3 - advanced respiratory support alone, or basic respiratory support together with support of at least two organ systems (includes all complex patients requiring support for multi-organ failure). Due to changes in the protocol, there were no subjects enrolled in the UK in Treatment Arm 4.
Time Frame: From Baseline up to Hospital Discharge
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 10 | 10 | 10 | 0
hour
  Level 0 and 1: number analyzed (Participants) | 9 | 10 | 9 | 0
  Level 0 and 1 | 74.64 (100.20) | 57.04 (40.36) | 64.39 (41.70) |
  Level 2: number analyzed (Participants) | 9 | 7 | 9 | 0
  Level 2 | 86.77 (45.84) | 62.34 (18.82) | 94.56 (84.96) |
  Level 3: number analyzed (Participants) | 0 | 1 | 2 | 0
  Level 3 |  | 66.80 | 14.10 (2.40) |

23. Secondary Outcome: Healthcare Resource Utilization: Team Managing the Participant During Hospitalization - Number of Healthcare Professional (HCP) Specialties Involved. (UK Participants Only)
Description: Number of Healthcare Professional (HCP) Specialists involved with care of participant during hospitalization of UK participants.Due to changes in the protocol, there were no subjects enrolled in the UK in Treatment Arm 4.
Time Frame: From Baseline up to Day 365
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: HCP per participant
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 10 | 10 | 10 | 0
HCP per participant | 3.9 (2.23) | 4.2 (1.93) | 4.0 (2.21) |

24. Secondary Outcome: Healthcare Resource Utilization: Number of Healthcare Professionals (HCP) Visits for Venous Thromboembolism (VTE) After Hospitalization and During 12month Follow-up. (UK Participants Only)
Description: Number of Healthcare Professional (HCP) Specialists involved with care of participant for Venous Thromboembolism (VTE) after hospitalization through 365 days for UK participants. Due to changes in the protocol, there were no subjects enrolled in the UK in Treatment Arm 4.
Time Frame: From Day 30 up to Day 365
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: HCP visits per participant
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 2 | 3 | 3 | 0
HCP visits per participant | 1.5 (0.71) | 1.3 (0.58) | 1.0 (0.00) |

25. Secondary Outcome: Healthcare Resource Utilization: Number of Healthcare Professionals (HCP) Visits for Venous Thromboembolism (VTE) After Hospitalization and During 12 Month Follow-up. (UK Participants Only)
Description: as for outcome 24
Time Frame: From Day 30 up to Day 365
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: HCP visits per participant
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 2 | 3 | 3 | 0
HCP visits per participant | 1.5 (0.71) | 1.3 (0.58) | 1.0 (0.00) |

26. Secondary Outcome: Healthcare Resource Utilization: Number of Hospital Re-Admissions After Hospitalization and During 12 Month Follow-up. (UK Participants Only)
Description: Number of Hospital Re-Admissions after hospitalization and during 12 month follow-up for UK Participants. Due to changes in the protocol, there were no subjects enrolled in the UK in Treatment Arm 4.
Time Frame: From Day 30 up to Day 365
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 0 | 0 | 1 | 0
Participants | 0 | 0 | 1 | 0

27. Secondary Outcome: Healthcare Resource Utilization: Duration of Hospital Re-Admissions After Hospitalization and During 12 Month Follow-up. (UK Participants Only)
Description: Duration of Hospital Re-Admissions after hospitalization and during 12 month follow-up for UK Participants. Due to changes in the protocol, there were no subjects enrolled in the UK in Treatment Arm 4.
Time Frame: From Day 30 through Day 365
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days per subject
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
Number analyzed (Participants) | 0 | 0 | 1 | 0
Days per subject |  |  | 2 (0) |

ADVERSE EVENTS:
Time Frame: From Baseline up to Day 365
Arm/Group | APT/2 Hours-r-tPA/2 mg/hr/Catheter | APT/4 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/1 mg/hr/Catheter | APT/6 Hours-r-tPA/2 mg/hr/Catheter
All-Cause Mortality (participants affected / at risk) | 1/37 | 1/37 | 0/37 | 1/18
Serious Adverse Events (participants affected / at risk) | 11/37 | 15/37 | 12/37 | 4/18
Other Adverse Events (participants affected / at risk) | 9/37 | 22/37 | 10/37 | 6/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | APT/2 Hours-r-tPA/2 mg/hr/Catheter (N=37) | APT/4 Hours-r-tPA/1 mg/hr/Catheter (N=37) | APT/6 Hours-r-tPA/1 mg/hr/Catheter (N=37) | APT/6 Hours-r-tPA/2 mg/hr/Catheter (N=18)
Aneamia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Anaemia postoperative (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 2
Fatigue (General disorders) | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 0 | 1 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Anticoagulation drug level below therapeutic (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0
Post thrombotic syndrome (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | APT/2 Hours-r-tPA/2 mg/hr/Catheter (N=37) | APT/4 Hours-r-tPA/1 mg/hr/Catheter (N=37) | APT/6 Hours-r-tPA/1 mg/hr/Catheter (N=37) | APT/6 Hours-r-tPA/2 mg/hr/Catheter (N=18)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 2
Anaemia postoperative (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac flutter (Cardiac disorders) | 0 | 1 | 0 | 0
Antithrombin III deficiency (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Chest pain (General disorders) | 2 | 1 | 1 | 2
Fatigue (General disorders) | 0 | 2 | 0 | 0
Gravitational oedema (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Vessel puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 3 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Coagulation factor VIII level increased (Investigations) | 0 | 0 | 1 | 0
Heart rate decreased (Investigations) | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental Status Changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 1 | 0
Postoperative renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Withdrawl bleed (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT02396758/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/58/NCT02396758/SAP_001.pdf